CLINICAL TRIAL: NCT06904443
Title: Effectiveness of a Temporal and Sound Space in the Paramedical Management of "Crisis" States of Patients Hospitalized in Psychiatry: Quasi-experimental Study With a Single Arm
Brief Title: Effectiveness of a Temporal and Sound Space in the Paramedical Management of "Crisis"
Acronym: PsySon
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: D23 P005
Record Dates: First submitted 2025-03-10; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-01

CONDITIONS: Psychiatric Hospitalization
MeSH Terms: interventions — Hospitals

STUDY DESIGN:
Intervention Model Description: Quasi-experimental efficacy study, using a historical control arm. The evaluation of the efficacy of the intervention will be carried out by comparing the results of the patients benefiting from the PSYSON device integrated into the nursing and paramedical monitoring with those of a historical cohort built from the GHU Health Data Warehouse (EDS) for the years 2022 and 2023, in the same departments participating in the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a historic control (No Intervention): a historical cohort constructed from the GHU Health Data Warehouse (EDS), including all patients meeting the inclusion/exclusion criteria, relating to the years 2022 and 2023, in the same departments participating in the study.
- psyson device (Experimental): during his hospitalization, the patient can benefit from listening sessions thanks to an original and innovative device, a sort of listening chair equipped with high-quality speakers, thus offering an immersive and enveloping experience (see photo). These sessions aim to anticipate or manage a moment of crisis, of "less well", which patients often face in institutions.
  Interventions: Other: PsySon is an innovative device that uses music in crisis management in hospitals

INTERVENTIONS:
Other: PsySon is an innovative device that uses music in crisis management in hospitals — during his hospitalization, the patient can benefit from listening sessions thanks to an original and innovative device, a sort of listening chair equipped with high-quality speakers, thus offering an immersive and enveloping experience (see photo). These sessions aim to anticipate or manage a moment of crisis, of "less well", which patients often face in institutions.
  Arms: psyson device

SUMMARY:
This project could potentially lead to better crisis management in psychiatry, using music as a mediator. The integration of a well-designed sound device could help caregivers build trust with patients, alleviate anxiety, and foster an environment conducive to healing. In addition, it would offer a less invasive and more patient-centered alternative, creating an atmosphere that facilitates communication and calming.

DETAILED DESCRIPTION:
The patient will receive specific, individualized paramedical monitoring. The PSYSON device will be presented to the patient during a paramedical interview within 3 days of the inclusion visit, by a pair of investigators composed of a nurse and a paramedic (occupational therapist or psychomotor therapist) or a psychologist.

This interview will help define the patient's personalized sound environment, adapted to moments of anxiety. The pair of investigators plays a key role in creating the playlist, which will constitute the patient's specific sound environment.

The first caregiver investigator will act as a close observer, observing the patient's reactions and psycho-corporal state, which could indicate psychomotor relaxation. The second caregiver investigator will use a tablet or computer provided by the department to enter the patient's choices into the application.

During this interview, the investigator will focus on the patient's emotions and sensory perception. It will begin with the patient's musical request, and to help the patient express his preferences, the investigator can rely on photo language, using "musical atmosphere" cards created for this purpose. These cards highlight a central musical theme, likely to arouse the patient's attention, emotion and certain ideas. Musical instruments can also be made available to observe the patient's musical and rhythmic desires and preferences.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 65 years old.
* Diagnosis of bipolar disorder or schizophrenia DSM5.
* Be hospitalized full-time in an acute psychiatric ward with or without compulsory care (SPL, SPDT, SPDTU, SPPI, SPDRE).
* Prior written informed consent of the patient or his legal representative.
* Benefit from a social protection scheme.

Exclusion Criteria:

* Have a severe cognitive disorder assessed during the clinical interview, making it impossible to focus one's attention.
* Hearing-impaired subjects who do not wear hearing aids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
administrations of conditional or emergency prescription medications for crisis conditions (states of stress, agitation, anxiety, etc.), during the first month of hospitalization for patients benefiting from the PSYSON system | 1 month
  change in the number of administrations of conditional or emergency prescription